CLINICAL TRIAL: NCT02007980
Title: Examining the Underlying Factors That Cause Ureteral Stent Discoloration in Japanese and Canadian Ureteral Stents
Brief Title: Indwelling Stent Discoloration Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver General Hospital (Other)
Responsible Party: Principal Investigator, Ben Chew, MD, Associate Professor, University of British Columbia
Other Study IDs: H13-02715
Record Dates: First submitted 2013-11-12; First posted 2013-12-11 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Urologic Injuries; Disorder of Urinary Stent; Kidney Calculi; Urinary Tract Obstruction Due to Specified Cause; Hydronephrosis
Keywords: urological problems; indwelling urologic stent; kidney stone disease; urinary system obstruction; hydronephrosis; ureteral damage
MeSH Terms: conditions — Kidney Calculi; Hydronephrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with indwelling ureteral stent: Patients with existing indwelling ureteral stent, no additional treatment

SUMMARY:
The aim of this study is to identify the root cause for the significant discolouration of Boston Scientific Percuflex based stents.

DETAILED DESCRIPTION:
The aim of this study is to identify the root cause for the significant discolouration of Boston Scientific Percuflex based stents observed in some patients, particularly those from Japan. We will also test and compare them to stents from Canadian patients. Furthermore, we will determine whether the discolouration promotes bacterial adhesion and/or encrustation of the stent.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 19 years of age (Vancouver, British Columbia, Canada - for Japan different age limit as applicable)
* Patient has indwelling ureteral stent

Exclusion Criteria:

* Pregnancy
* Positive Urine Culture
* Active cancer
* Recurrent urinary infections
* Gross hematuria
* Inability to provide informed consent
* Physician/Surgeon refuses to enter patient into study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with indwelling ureteral stent due to urologic indication.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
stent encrustation | at stent removal
  Conditioning film components and encrustation

SECONDARY OUTCOMES:
characterize the components that discolour the Percuflex material | bench top testing of stents
Bacterial Adhesion, Colonization, and Biofilm formation | at 4, 24, and 48 hours post stent removal
  Stent pieces from the stent that has been in the patient will be exposed to bacteria and artificial urine to mimic ureter environment in order to find information on: bacterial adhesion, colonization and biofilm formation

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — UBC/VGH
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada